CLINICAL TRIAL: NCT03390569
Title: Does Exercise Improve Progression-free Survival in Glioblastoma? A Prospective Single Arm Intervention Trial
Brief Title: Exercise in Patients With Glioblastoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); University of Toronto (Other); McMaster University (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-5922
Record Dates: First submitted 2017-09-27; First posted 2018-01-04 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Glioblastoma
Keywords: GBM; Glioblastoma; Brain Cancer; High-Grade Glioma; Glioma
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Glioma | interventions — Exercise; Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise in GBM (Experimental): All patients will be assigned a three-month exercise intervention according to their own capabilities and current activity levels
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — The patients meet with a registered physiotherapist and receive individualized exercise programs starting the second week of treatment, and continuing up to 3 months later.
  Other Names: Fitness; Physiotherapy

SUMMARY:
Patients with newly-diagnosed GBM will be given personalized exercise regimes during concurrent chemo-radiation and up to 3 months later. Study aims are to investigate the feasibility and preliminary efficacy of the exercise program on progression free survival. Secondary outcomes of interest include cognition, fatigue, and quality of life.

DETAILED DESCRIPTION:
Background: Glioblastoma (GBM) is the most common malignant glioma in adults, with a very poor prognosis, limited new treatment options, and neurological sequelae, including physical and cognitive decline that adversely affect quality of life (QOL). Physical activity may be an intervention that attenuates the cognitive and physical decline associated with GBM. However, few studies examine physical activity in brain tumor patients, perhaps due to challenges in trial design, measuring outcomes, and complexity of care. Aims of this work are to develop and implement an individualized exercise intervention for GBM patients to support functional independence, and to delay tumor progression and cognitive decline. Methods: GBM patients scheduled to be treated with concurrent radiation and chemotherapy will be recruited from the neuro-oncology clinic at the Princess Margaret Cancer Centre. Participants will receive an individualized, home-based exercise program that includes aerobic and resistance training, tailored to prior level of fitness, current physical status, and individual interests. They will undergo 1-hr standardized, validated assessments of physical and neurocognitive functions, mood, fatigue, and QOL, prior to radiation, and then 3, 6, 12, and 18 months later. Significance: Identifying interventions that preserve or improve mobility and cognitive function will enhance QOL and may lengthen progression-free survival in brain tumor patients. Moreover, finding ways to help patients maintain self-care will lessen the strain on the health care system (e.g., fewer hospitalizations, delayed utilization of palliative care hospice).

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed glioblastoma
* fluent in English
* scheduled to be treated with concurrent chemoradiation (or within 2 weeks of starting treatment)

Exclusion Criteria:

* brain metastases secondary to non-central nervous system cancer
* less than 18 years old
* receiving treatment at a location other than the Princess Margaret Cancer Centre
* deemed unfit to exercise by a study oncologist
* lack of fluency in English
* psychiatric or neurological disorders that could interfere with participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | 6 months
  Time to tumor progression, based on Response Assessment in Neuro-Oncology (RANO) criteria

SECONDARY OUTCOMES:
Cognitive Decline | 3 months, 6 months, 12 months, 18 months post-treatment
  Tests will be scored according to published criteria, converted to z-scores based on population norms, and averaged to create an overall cognitive function score. COgnitive decline will be defined as declined scores at a given time point (preservation of cognitive functions will be defined as stable or improved scores at a given time point).
Cognitive Complaints | 3 months, 6 months, 12 months, 18 months post-treatment
  as measured by a validated questionnaire
Overall survival | Up to 18 months post-treatment
  rate of overall survival
Personality Changes | 3, 6, 12 and 18 months post-treatment
  as measured by a standardized questionnaire
Quality of Life | 3, 6, 12 and 18 months post-treatment
  as measured by a validated questionnaire
Mood | 3, 6, 12 and 18 months post-treatment
  as measured by a validated questionnaire
Interference with valued activities and interests | 3, 6, 12 and 18 months post-treatment
  as measured by a validated questionnaire
Sleep Quality | 3, 6, 12 and 18 months post-treatment
  as measured by a validated questionnaire
Physical Function | 3, 6, 12 and 18 months post-treatment
  strength, balance, cardiovascular endurance

CONTACTS AND LOCATIONS:
Overall Officials: Kim Edelstein, PhD, C.Psych., Principal Investigator — University of Toronto, University Health Network; Warren Mason, MD, Principal Investigator — University of Toronto, University Health Network; Kristin Campbell, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Princess Margaret Hospital, University Health Network, Toronto, Ontario, Canada